CLINICAL TRIAL: NCT03108508
Title: Randomized, Crossover, Double Blinded, Non-inferiority Study of Three Products Rich in Organic Silicon, in Postprandrial Situation
Brief Title: Non-inferiority Bioavailabilty Study of 3 Silicon-rich Supplements
Acronym: BIOSILICI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technological Centre of Nutrition and Health, Spain (Other)
Collaborators: SILICIUM ESPAÑA LABORATORIOS SLU (Unknown); Hospital Universitari Sant Joan de Reus (Other); University Rovira i Virgili (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: BIOSILICI
Record Dates: First submitted 2017-03-29; First posted 2017-04-11 (Actual); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: Absorption; Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Prod1 (Experimental): G5 Siliplant
  Interventions: Dietary Supplement: Prod1
- Prod2 (Experimental): Orgono Powder®
  Interventions: Dietary Supplement: Prod2
- Prod3 (Experimental): G7 ALOE
  Interventions: Dietary Supplement: Prod3

INTERVENTIONS:
Dietary Supplement: Prod1 — 60 mL of product (water, silicic acid, Equisetum Arvense, Rosmarinus officinalis) (Silicic acid) equivalent to 21.6 mg of elemental silicon.
  Other Names: G5
  Arms: Prod1
Dietary Supplement: Prod2 — 1.4 g of product (Orthosalicic acid) equivalent to 21.6 mg of elemental silicon
  Other Names: Orgono powder
  Arms: Prod2
Dietary Supplement: Prod3 — 120 mL of product (Aloe barbadensis Miller, organic silicon, potassium sorbate, cítric acid) (Organic silicon) equivalent to 21.6 mg of elemental silicon
  Other Names: G7 Aloe
  Arms: Prod3

SUMMARY:
The objective of the present study is to evaluate the non-inferiority of the absorption parameters of three silicon supplements in human volunteers.

DETAILED DESCRIPTION:
The objective of the present study is to evaluate the non-inferiority of the absorption parameters of three silicon supplements in human volunteers.

Participants: 5 healthy men over 18 years old, with normal serum creatinine levels. Treatment consists of one product consumption every week, and measuring postprandrial response at 0, 30, 60, 90, 120, 180, 240 and 360 min, in blood, and urine in two periods of three hours each.

The statistical analysis will follow the principles specified in the guidelines of the ICHE and CPMP/EWP/908/99 ICHE Points to Consider on Multiplicity Issues in Clinical Trials.

ELIGIBILITY:
Inclusion Criteria:

* Adults men or women (>18 years old)
* With normal serum creatinine levels.
* Written informed consent provided before the initial screening visit.

Exclusion Criteria:

* Suffering from chronic diseases
* Suffering from intestinal disorders
* Consuming silicon supplements in the 7 days prior to inclusion in the study.
* Consuming medicines containing silicon in the 7 days prior to inclusion in the study.
* Current or past participation in a clinical trial or consumption of a research product in the 30 days prior to inclusion in the study.
* Failing to follow study guidelines.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-07-30 (Actual)

PRIMARY OUTCOMES:
concentration of sillicium in urine samples | Urine will be collected in two 3-h collections (0-180min and 181-360 min) in two separate containers at Visit 1, Visit 2 and Visit 3 (1 week between visits)
  concentration of sillicium in urine samples will be measured by inductively coupled plasma optical emission spectrometry.

SECONDARY OUTCOMES:
concentration of sillicium in plasma | Blood samples will be collected to determine baseline plasma silicon value (time 0 min = T0). After ingestion of one of the study products, additional blood samples will be collected at 30, 60, 90 and 120 min at Visit 1, Visit 2 and Visit 3
  concentration of silicon in blood/plasma samples will be measured by inductively coupled plasma optical emission spectrometry.
  .

CONTACTS AND LOCATIONS:
Locations (1):
- Technological Centre of Nutrition and Health (CTNS), Reus, Tarragona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Technological Centre of Nutrition and Health — http://www.ctns.cat/en